CLINICAL TRIAL: NCT00706251
Title: Long Term Follow up of Nasolacrimal Intubation in Adults With Mild Epiphora
Brief Title: Follow up of Nasolacrimal Intubation in Adults
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Arie Nemet, MD, Shaare Zedek Medical center, Maccabi Healthcare Services
Other Study IDs: LTFNIAME
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Lacrimal Apparatus Diseases; Dacryocystitis
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Dacryocystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary: All the patients in our medical center who underwent nasolacrimal intubation, due to mild epiphora, during the years 2000-2007.
  Interventions: Device: Silicone tube

INTERVENTIONS:
Device: Silicone tube — Silicone tube which is inserted into the tear duct through the punctum in the eyelid, then passed through the tear duct till it enters the nose and secured in place using a surgical knot. The tube remains in place for 3-6 months, than take out by the surgeon.

SUMMARY:
For patients with chronic epiphora, Dacryocystorhinostomy is currently the gold standard treatment, with a success rate of 80-90% according to literature. Another available treatment, which is far less used, in nasolacrimal intubation, using a silicone tube.

In our study, we would like to find the efficacy of nasolacrimal duct intubation, which was performed in our medical center on a few hundred patients with mild epiphora.

Study hypothesis: nasolacrimal intubation in adults, with a clinically mild epiphora, is close in it's efficacy to the Dacryocystorhinostomy procedure.

DETAILED DESCRIPTION:
Under normal conditions, the amount of tears excreted from lacrimal glands to the eye is equal to the amount drained through the tear duct. Epiphora in adults usually involves a blockage of the lacrimal sac or the nasolacrimal duct. Epiphora causes tearing in patients, which can be treated sympthomatically in a conservative way (antibiotic treatment, probing of the tear duct, pressure irrigation of the tear duct) or therapeutic in an invasive way. The invasive treatment includes one of the following:

1. Dacryocystorhinostomy - surgery for reconstructing an alternative path for tear drainage.
2. Nasolacrimal intubation - inserting a silicone tube through the tear duct. The tube is usually removed after 3-6 months.

Currently, there are only a few reports regarding the efficacy of nasolacrimal intubation, all with a small number of research subjects. Also, these reports have stratified the patients according to the location of the tear duct blockage, and didn't take into account the severity of the blockage (ie the severity of symptoms) prior to performing the intubation.

In our research, we would like to find the efficacy of nasolacrimal intubation which was performed in our medical center on a few hundred patients with mild epiphora, and to compare in with the efficacy of the Dacryocystorhinostomy - which is 80-90% according to literature.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild epiphora.
* Underwent nasolacrimal intubation during 01/2000 - 12/2007.

Exclusion Criteria:

* Purulent excretions from nasolacrimal duct on day of admission or intubation.
* Nasolacrimal intubation in the past.
* Dacryocystorhinostomy in the past.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent nasolacrimal intubation in Maccabi Healthcare, due to mild epiphora, during the years 2000-2007.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2000-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Patient being completely free of tearing. | 1 year.

SECONDARY OUTCOMES:
Following nasolacrimal intubation, did the patient need a Dacryocystorhinostomy surgery. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arie Nemet, MD, Study Director — Shaare Zedek Medical Center, Maccabi Healthcare; Arie Nemet, MD, Study Chair — Shaare Zedek Medical Center, Maccabi Healthcare; Arie Nemet, MD, Principal Investigator — Shaare Zedek Medical Center, Maccabi Healthcare
Locations (1):
- Maccabi Healthcare Eye Clinic, Tel Aviv, Israel

REFERENCES:
- [Background] Becker BB, Berry FD, Koller H. Balloon catheter dilatation for treatment of congenital nasolacrimal duct obstruction. Am J Ophthalmol. 1996 Mar;121(3):304-9. doi: 10.1016/s0002-9394(14)70279-x. PMID 8597274
- [Background] Hurwitz JJ, Rutherford S. Computerized survey of lacrimal surgery patients. Ophthalmology. 1986 Jan;93(1):14-9. doi: 10.1016/s0161-6420(86)33779-5. PMID 3951812
- [Background] Keith CG. Intubation of the lacrimal passages. Am J Ophthalmol. 1968 Jan;65(1):70-4. doi: 10.1016/0002-9394(68)91031-3. No abstract available. PMID 5635571
- [Background] Quickert MH, Dryden RM. Probes for intubation in lacrimal drainage. Trans Am Acad Ophthalmol Otolaryngol. 1970 Mar-Apr;74(2):431-3. No abstract available. PMID 5445947
- [Background] Crawford JS. Intubation of obstructions in the lacrimal system. Can J Ophthalmol. 1977 Oct;12(4):289-92. PMID 922571
- [Background] Pashby RC, Rathbun JE. Silicone tube intubation of the lacrimal drainage system. Arch Ophthalmol. 1979 Jul;97(7):1318-22. doi: 10.1001/archopht.1979.01020020060014. PMID 454271
- [Background] Connell PP, Fulcher TP, Chacko E, O' Connor MJ, Moriarty P. Long term follow up of nasolacrimal intubation in adults. Br J Ophthalmol. 2006 Apr;90(4):435-6. doi: 10.1136/bjo.2005.084590. PMID 16547322